CLINICAL TRIAL: NCT03402282
Title: Upper Rectal Artery Embolization in the Treatment of Hemorrhoidal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 72364117.0.1001.0071
Record Dates: First submitted 2017-12-18; First posted 2018-01-18 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-08

CONDITIONS: Hemorrhoidal Disease
Keywords: hemorrhoidal disease; embolization
MeSH Terms: interventions — Embolization, Therapeutic; Wound Healing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- embolization (Experimental): upper rectal artery embolization
  Interventions: Procedure: embolization
- surgical treatment (Active Comparator): surgical repair through the classic technique (Milligan and Morgan technique)
  Interventions: Procedure: surgical repair

INTERVENTIONS:
Procedure: embolization — upper rectal artery embolization with coils
  Other Names: upper rectal artery embolization
  Arms: embolization
Procedure: surgical repair — surgical repair through the classic technique (Milligan and Morgan technique)
  Arms: surgical treatment

SUMMARY:
Hemorrhoidal disease diagnosis is based on medical history combined with physical exam and complementary exam. Physical exam should include inspection at exertion, digital rectal exam ,and anoscopy.

The treatment indicated in patients with hemorrhoidal disease varies according to the disease grade, and it may be clinical or surgical. The classic surgical approach is an open surgical correction , a technique that has high success rates and low recurrence rates; however, it is accompanied by intense pain.

Based on the concept that hemorrhoids are formed by pathological changes in submucosal pads vascularization in anal channel transition zone, selective embolization of upper rectal artery branches were performed in 14 patients with long-term severe rectal bleeding secondary to hemorrhoidal disease by Vidal et al. with no pain or ischemic symptoms being seen.

* Main Objective To determine the feasibility of implementing upper rectal artery embolization in the treatment of patients with grade 2 (protrude beyond the anal verge with straining or defecating but reduce spontaneously) and 3 hemorrhoids (protrude spontaneously or with straining and require manual reduction), relating its short- and long-term outcomes with patients undergoing surgical repair through the classic technique
* Hypothesis The expectation is that, with upper rectal artery embolization, patients experience a decrease or remission of symptoms, such as bleeding, pain and symptoms related to hemorrhoidal pads edema. Another expectation is that the decrease in the number of days to return to daily activities

DETAILED DESCRIPTION:
Proposal description 1.1. Hemorrhoids: Epidemiology, Clinical Presentation and Diagnostic Assessment: In the normal anal channel, there are three highly-vascularized areas (pads), forming slight masses in the submucosa made of blood vessels, smooth muscle and elastic and connective tissue, and are located at the left lateral, right anterior and right posterior quadrants, and contribute in anal continence . The term hemorrhoids refers to clinical situations where these hypervascularized pads are abnormal and cause clinical symptoms.

The exact disease prevalence of symptomatic hemorrhoidal disease is difficult to establish, since many symptomatic patients do not seek an assessment, while others assign varied anorectal symptoms as being resulting from hemorrhoids. Some series estimate prevalence between 4 and 40 %. Although many patients will exhibit symptomatic hemorrhoids along life, the peak incidence occurs between 45 and 65 years old and its development prior to 20 years old is rarely frequent . Among the factors related to a higher risk of developing the disease are: pregnancy, white race, females.

Hemorrhoids may be divided as external and internal. External hemorrhoids are covered by anoderm (richly enervated layer), are located distally to the dentate line and their main symptoms are edema, causing discomfort and difficult local hygiene, which may also exhibit an intense pain when thrombosed. Internal hemorrhoids are located proximally to the dentate line and are lined with poorly enervated anorectal mucosa, and rarely cause pain, except when thrombosed and combined with prolapse and necrosis; often their symptoms are prolapse and bleeding.

Internal hemorrhoids may be subdivided into 4 grades: grade 1 are defined by a protuberance in anal channel and may show prolapse beyond the dentate line at great exertion; grade 2 are hemorrhoids prolapsing beyond the dentate line at exertion, but reduced spontaneously; grade 3 are hemorrhoids prolapsing beyond the dentate line, requiring manual reduction; and grade 4 are defined by non-reducing prolapsed hemorrhoids, being at risk of strangulation.

Hemorrhoidal disease diagnosis is based on medical history combined with physical exam and complementary exam. Physical exam should include inspection at exertion, digital rectal exam (which allows an assessment of internal and external hemorrhoids, anal channel tonus assessment, in addition to excluding other diseases, such as neoplasm and sphincter spasm) and anoscopy. Among complementary tests, flexible rectal sigmoidoscopy, colonoscopy, barium enema may be requested at complementary diagnosis, mainly to rule out other diseases.

1.2. Hemorrhoids: conventional treatment: non-surgical and surgical

The treatment indicated in patients with hemorrhoidal disease varies according to the disease grade, and it may be clinical or surgical. Non-surgical management is indicated for patients with internal and external hemorrhoids (grade 1 to 4) and consists in better local hygiene, avoiding excessive exertion and improving food habits (including more fibers in the diet), combined or not with laxative drugs. Patients with prolapsed external or internal hemorrhoids may further benefit from the combination of clinical measures and more invasive measures such as rubber band ligation, sclerotherapy and electrocoagulation.

Surgical management is best indicated in patients failing clinical measures and patients with grade 3 and 4 hemorrhoids, and is indicated in about 10% of cases . The classic surgical approach is an open surgical correction through Milligan and Morgan technique, which comprised resection and ligation as high as possible of the three arterial pedicles feeding the hemorrhoids, a technique that has high success rates and low recurrence rates; however, it is accompanied by intense pain ( with pain scale in the first 24 hours of approximately 6.1 ± 1.5; in the first evacuation 4.5 ± 1.5) and a prolonged recovery period to return to normal activities (6.95 ± 3.6 days). Currently, two less invasive new techniques with less intense post-operative pain were proposed: anopexy with circular stapler (Longo's technique- which consists of interrupting the superior rectal branches and resecting the rectal mucosal ring, it is less invasive, but not free from complications which may range from urinary retention (1.9 to 5%) rectal-vaginal fistulae, bleedings requiring blood transfusion (1.5 a 9%), external hemorrhoidal thrombosis (1.2 a 4.7%) and perforations) and Doppler-guided elective ligation of hemorrhoidal artery through endoanal access ; however, these have a recurrence higher than 10% and complications from 6 to 22% of cases such as: bleeding, urinary retention, hematoma in the submucosa, fissure, abscess. Both techniques are associated with reduction of arterial flow with subsequent reduction of hemorrhoids .

1.3. Hemorrhoids: Hemorrhoidal Artery Embolization

Based on the concept that hemorrhoids are formed by pathological changes in submucosal pads vascularization in anal channel transition zone, Galkin in 1994 reported the first cases of treating hemorrhoidal disease through embolization of upper hemorrhoidal branches in 34 patients, without recurrence after 24 months of follow-up.

Recently, Vidal et al 2014 describe the "emborrhoid" technique, consisting in super selective embolization of upper rectal artery branches. "Emborrhoid" technique was performed through right common femoral artery puncture (inserting a 5Fr introducer) and catheterization of lower mesenteric artery with a Simmons catheter, followed by a super selective catheterization of lower rectal arteries with a microcatheter and embolization with Nester 0.018 coils with 2 and 3 mm of diameter and 3-cm long. This technique was performed in 14 patients with long-term severe rectal bleeding secondary to hemorrhoidal disease grades 2 (10 patients), 3 (3 patients) and 4 (1 patient) who were not candidates to other clinical or surgical therapies after a multidisciplinary discussion . The technical success was seen in a 100% of cases. After a follow-up between 2 and 13 months, clinical success (no bleeding or minimum bleeding and well tolerated by the patient) occurred in 72% (10/14) of cases, with no pain or ischemic symptoms being seen. Four patients experienced new bleeding, of these, 2 underwent a new embolization and 2 refused further treatment.

Moussa et al performed upper rectal arteries embolization with the "emborrhoid" technique described by Vidal et al in 30 patients with hemorrhoidal disease and an immediate technical success was observed in 93% of cases, with no pain in the postoperative period and absence of complications related to puncture site or ischemic, such as rectal ulceration, anal fissure.

1.3.1. Complications Related to Conventional Surgical Treatment The possible early complications related to conventional surgical treatments are pain, urinary retention (2-36%), intestinal constipation, bleeding (0.03- 6%) and infection (0.5-5.5%). And the late complications may include anal incontinence (flatulence and / or stools- 2-12%) and anal stenosis (0-6%).

1.3.2 Complications Related to Upper Rectal Artery Embolization: The possible complications related to upper rectal artery embolization relate to the puncture site and potential rectal ischemia. However, with the use of coils, this risk is decreased, since it does not cause distal embolization, as per Vidal et al, who reported 14 cases of coil embolization at upper rectal arteries, with no rectal ischemia symptoms seen.

2. Study Objectives: Main Objective To determine the feasibility of implementing upper rectal artery embolization in the treatment of patients with grade 2 (protrude beyond the anal verge with straining or defecating but reduce spontaneously) and 3 hemorrhoids (protrude spontaneously or with straining and require manual reduction), relating its short- and long-term outcomes with patients undergoing surgical repair through the classic technique (Milligan and Morgan technique).

Hypothesis The expectation is that, with upper rectal artery embolization, patients experience a decrease or remission of symptoms, such as bleeding, pain and symptoms related to hemorrhoidal pads edema. Another expectation is that the decrease in the number of days to return to daily activities.

3. Materials and Methods This project will be developed by using the "Emborrhoid" technique described by Vidal et al. , consisting in upper rectal artery embolization with coils for patients with hemorrhoidal disease exhibiting chronic bleeding, and it has been shown to be safe and efficient .

This research project will be developed together with the Hospital Israelita Albert Einstein - Morumbi Unit and the Vila Santa Catarina Municipal Hospital, with patients recruited from grade 2 and 3 hemorrhoidal disease patients requiring surgical treatment referred to Hospital Vila Santa Catarina-Hospital Israelita Albert Einstein who accept to take part in the research protocol. Patients will undergo a detailed clinical and proctological evaluation, in addition to colonoscopy, and will then be assigned to 2 groups with 20 patients each (embolization or conventional surgical treatment groups) in a random way. Patients assigned to embolization group will be referred to the hemodynamics department of Hospital Israelita Albert Einstein - Morumbi Unit to undergo upper hemorrhoidal artery embolization, by an experienced interventional radiology team (>5 years of experience) and patients assigned to conventional surgical treatment group will be treated at Hospital Vila Santa Catarina by an experienced proctologists team (> 10 years of experience).

Follow-up will be performed with visits at post-operative days 7 and 30 , as well as telephone calls at 1, 3, 6, and 12 months. Patients will fill out a questionnaire at home during the first week, to evaluate their pain symptoms through the Visual Analogue Scale, at the following moments: first evacuation, first and third days, and report the number and number of times it was necessary to use analgesic and/or anti-inflammatory medication.

3.2. Inclusion Criteria Male and female patients aged above 18 years old, with internal and/or external hemorrhoids experiencing clinical symptoms (anemia, persistent / recurrent bleeding hemorrhoidal source> 3 months, episodes of recurrent hemorrhoidal thrombosis (> 2 episodes) or associated the symptoms of hemorrhoidal disease) with surgical indication and contraindication of band ligation and / or photocoagulation infrared accepting the items pointed in the informed consent form.

3.3. Exclusion Criteria Patients with contraindications for angiogram performance (allergy to intravenous contrast), patients with aortic atherosclerosis (femoral pulse and difference Doppler angiography or with stenosis 20%) patients in the daily use of NSAIDs or weak opioids or who refuse to take part in this project will be excluded from this study.

3.4. Study Dynamics Patients from conventional surgical treatment group will undergo the standard treatment for hemorrhoidal disease at Hospital Vila Santa Catarina and patients from embolization group will be referred to Hospital Israelita Albert Einstein, where they will undergo pelvic angiogram, assessing possible anatomical variations, followed by a super selective catheterization of upper rectal artery branches and coil embolization of these branches, followed by a controlled pelvic angiography and compression for 30 minutes of the puncture site after the end of the procedure. After the procedure, the rates of technical success and early and intermediate-term clinical success will be assessed, as well as potential complications.

3.5. Sample Calculation Based on the literature, the expected value of pain given by the visual analogue scale on the first 10 days of surgery was 4.2 in patients submitted to hemorrhoidectomy using the classic Milligan-Morgan technique, with the variability of 2.24 (DP = 2,24 pontos) . It is expected patients who underwent the procedure present a maximum of 2 points at pain scale in the same period. With an 80% of power and 95% confidence - it's only required 20 subjects for the study.

3.6. Randomization Allocation of patients in the 2 groups will be performed through randomization, in blocks consisting of 4 individuals in each block, in order to reduce the variability and potential confounding between the 2 groups.

4. Informed Consent

All patients should be given informed consents

5. Ethical Considerations 5.1. Declaration of Helsinki

The participating researcher will ensure that this program will be conducted in full compliance with the Helsinki Declaration and all local and national regulations.

5.2. Safety

5.2.1 Adverse Events and Complications Graduation Criteria Adverse events and complications were classified according to the terminology criteria of the National Institutes of Health (NIH) (4.0; edition 28.05.2009 version).

5.2.2. DSMB - Data Safety Monitoring Board The primary safety result of the study (local complications of puncture site and rectal ischemia) will be reviewed by an independent Data Safety Monitoring Board, composed of at least one general surgeon / proctologist and one interventional vascular radiologist. In locu analyzes will be performed at every 10 patients submitted to treatment (according to the randomization of the groups). The meeting will be programmed according to the recruitment and will be schedule with the inclusion of 1/4, 1/2, 3/4 of the participants (10 participants, 20 participants, 30 participants respectively)

6. Confidentiality of data The team involved in the study pledges to keep under confidentiality all the information here displayed as well as use the data only for the specific purposes of this study.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged above 18 years old, with internal and/or external hemorrhoids experiencing clinical symptoms (anemia, persistent / recurrent bleeding hemorrhoidal source> 3 months, episodes of recurrent hemorrhoidal thrombosis (> 2 episodes) or associated the symptoms of hemorrhoidal disease) with surgical indication and contraindication of band ligation and / or photocoagulation infrared accepting the items pointed in the informed consent form.

Exclusion Criteria:

* Patients with contraindications for angiogram performance (allergy to intravenous contrast), patients with aortic atherosclerosis (femoral pulse and difference Doppler angiography or with stenosis 20%) patients in the daily use of NSAIDs or weak opioids or who refuse to take part in this project will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
short and long upper rectal artery versus surgical repair the classic technique | 1.5 years
  To determine the feasibility of implementing upper rectal artery embolization in the treatment of patients with grade 2 (protrude beyond the anal verge with straining or defecating but reduce spontaneously) and 3 hemorrhoids (protrude spontaneously or with straining and require manual reduction), relating its short- and long-term outcomes with patients undergoing surgical repair through the classic technique (Milligan and Morgan technique).

SECONDARY OUTCOMES:
impact of upper rectal artery embolization on the treatment of hemorrhoidal disease | 1.5 years
  To assess the impact of upper rectal artery embolization on the treatment of chronic bleeding secondary to hemorrhoidal disease, on clinical success rate.
clinical success of upper rectal artery embolization on the treatment of hemorrhoidal disease. | 1.5 years
  To assess the impact of upper rectal artery embolization on the treatment of chronic bleeding secondary to hemorrhoidal disease, on need of retreatment.
improves symptoms | 1.5 years
  To assess the impact of upper rectal artery embolization on the treatment of chronic bleeding secondary to hemorrhoidal disease, on symptom relapse
clinical recovery | 1.5 years
  To assess the impact of embolization on the time required for clinical recovery and return to daily activities
Pharmacoeconomic | 1.5 years
  Pharmacoeconomic assessment of the comparison between upper rectal artery embolization methods for hemorrhoidal disease treatment and conventional surgical treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, Brazil

REFERENCES:
- [Derived] Falsarella PM, Katz M, Affonso BB, Galastri FL, Arcuri MF, Motta-Leal-Filho JMD, Araujo SEA, Garcia RG, Nasser F. Angiographic description of the superior rectal artery and its anatomical variations in patients undergoing embolization of the superior rectal arteries in hemorrhoidal disease treatment. Einstein (Sao Paulo). 2024 Sep 30;22:eAO0688. doi: 10.31744/einstein_journal/2024AO0688. eCollection 2024. PMID 39356943